CLINICAL TRIAL: NCT03508427
Title: Toi Même: a Mobile System for Measuring Bipolar Illness Activity - Feasibility Study
Brief Title: Toi Même: a Mobile System for Measuring Bipolar Illness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended since april 2020 as the application is temporarily unavailable
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-004
Record Dates: First submitted 2017-11-17; First posted 2018-04-25 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Smartphone; Self-monitoring; Objective data
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: One-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toi Même plus treatment as usual (Experimental): One-Arm study Intervention: Toi Même self-monitoring smartphone application plus treatment as usual which includes pharmacological and/or psychological treatment.
  Tool: Toi Même mobile app
  Interventions: Other: Daily self-monitoring

INTERVENTIONS:
Other: Daily self-monitoring — Toi Même self-monitoring smartphone application plus treatment as usual which includes pharmacological and/or psychological treatment.

SUMMARY:
Bipolar disorder is a severe psychiatric illness with chronic course and it is associated with high risk of relapse and hospitalisation, and many patients do not recover to their previous psychosocial functioning. Major reasons for poor outcomes are delayed intervention for prodromal mood and behavioural symptoms as well as incomplete treatment responses. Current diagnostic approaches used to assess mood symptoms rely on symptom-based categories, which lack sensitivity to detect subtle mood and behavioural changes. Therefore, the ability to better characterizing bipolar patients may allow to detect possible differences in the illness activity.

On the other hand, there is a growing interest in the potential use of mobile technologies such as mobile apps, smartphone and internet in psychiatric care. Some projects have been testing the potential benefits of mobile apps to assess and treat individuals at-risk or suffering from mood and bipolar disorders, using online signs and symptoms monitoring, yet to the investigators knowledge, none of them have integrated a dimensional approach in a smartphone app to assess mood and behavioural alterations and bipolar illness activity, including subjective and objective data (e.g. physical activity, social activity, etc.).

In this feasibility study the investigators will evaluate the potential relevance of Toi Même app to self-monitoring mood and behavioural changes in bipolar patients with different mood phases compared to the gold-standard mood rating tools used in clinical practice. All patients will be followed for 3 months, with outcome assessments after 2 weeks, after 1 month, 2 months and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with the current diagnosis of Bipolar disorder type I or type II according to the DSM-5 criteria
* having an iPhone with iOS version from 9.x with access to wireless Internet connectivity.

Exclusion Criteria:

* Current DSM-5 diagnosis of schizophrenia, psychotic disorders, dementia, or mental retardation.
* Active suicidal ideation or behaviours.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Severity of depressive symptoms | 3 months study period
  Changes in depressive symptoms measured using the Montgomery-Asberg Depression Rating Scale during the 3 months study period.
Severity of manic symptoms | 3 months study period
  Changes in manic symptoms measured using the Young Mania Rating Scale during the 3 months study period.

SECONDARY OUTCOMES:
Self-rated depressive symptoms | 3 months study period
  Differences in self-rated depressive symptom using the Quick Inventory of Depressive Symptomatology (QIDS) during the 3 months study period.
Self-rated manic symptoms | 3 months study period
  Differences in self-rated manic symptoms using the Altman Mania Self-Rating Scale (ASRM) during the 3 months study period.
Activation levels | 3 months study period
  Changes in levels of activation measured using the scale Multidimensional Assessment of Thymic States (MAThyS) during the 3 months study period.
Treatment adherence | 3 months study period
  Differences in treatment adherence using the 10-item Medication Adherence Rating Scale (MARS) during the 3 months study period.
Functional impairment | 3 months study period
  Differences in functional impairment using the Functioning Assessment Short Test (FAST) during the 3 months study period.
Movement behavior | 3 months study period.
  Differences in movement behavior using the smartphone motion sensors during the 3 months study period.
Completion rate | 3 months study period.
  Differences in the completion rate of app self-assessment questionnaires.
Patient acceptance | 3 months study period.
  Patient acceptance rate measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Henry, MD PhD, Principal Investigator — Institut Pasteur
Locations (3):
- France (3):
  - Nightingale Hospitals Paris - Clinique du Château, Garche
  - Centre Thérapeutique et Preventif de Jour - Troubles Bipolaires (Clinique Bellevue), Meudon, Île-de-France Region
  - Centre Hospitalier Sainte Anne, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dargel AA, Mosconi E, Masson M, Plaze M, Taieb F, Von Platen C, Buivan TP, Pouleriguen G, Sanchez M, Fournier S, Lledo PM, Henry C. Toi Meme, a Mobile Health Platform for Measuring Bipolar Illness Activity: Protocol for a Feasibility Study. JMIR Res Protoc. 2020 Aug 18;9(8):e18818. doi: 10.2196/18818. PMID 32638703